CLINICAL TRIAL: NCT04260880
Title: Assessment of Periodontal Status in Patients With Depression : A Cross Sectional Study.
Brief Title: Periodontal Assessment in Depression Patients
Status: Completed | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: APARNA PGIDS/IEC/2019/31
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Periodontitis; Depression
MeSH Terms: conditions — Periodontitis; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Test group 1: individuals with mild depression
  Interventions: Other: periodontal status in mild depression patients
- Test group 2: individuals with moderate depression
  Interventions: Other: periodontal status in moderate depression patients
- control group: systemically healthy individuals
  Interventions: Other: periodontal status in systemically healthy patients

INTERVENTIONS:
Other: periodontal status in mild depression patients — Assessment of periodontal status in mild depression patients
  Groups: Test group 1
Other: periodontal status in moderate depression patients — Assessment of periodontal status in moderate depression patients
  Groups: Test group 2
Other: periodontal status in systemically healthy patients — Assessment of periodontal status in systemically healthy patients
  Groups: control group

SUMMARY:
To assess the periodontal status in the patients with depression. Evaluation of periodontal status in patients with mild depression. Evaluation of periodontal status in patients with moderate depression. Evaluation of periodontal parameters in patients without depression.

DETAILED DESCRIPTION:
Periodontitis, a periodontal disease, results from interaction between the immune system and oral bacteria that may promote oxidative stress and initiate an inflammatory cascade inducing the destruction of the oral structure.

The immune-microbial pathogenesis of periodontitis involves chronic inflammation, which alters the balance among multiple systems, including the neural, immune, and endocrine systems. Multiple systemic conditions, such as diabetes, cardiovascular diseases, and respiratory diseases, have been shown to have an inflammatory association with periodontitis, and pro-inflammatory cytokines such as tumor necrosis factor (TNF)-a, interleukin (IL)-1, and IL-6 are involved. In addition, distress experienced by the patients with periodontitis showed correlation with the progression of periodontitis. Studies have demonstrated that chronic stress and depression fall into a spectrum and could induce dysregulation of the immune system, impairing the course of periodontitis.

Depression, a disabling psychiatric disorder, manifests with depressed mood, vegetative symptoms, and cognitive impairment, and could impair the personal life quality and physical function. In 2015, this mental disorder was classified as the third main cause of global disability . It is a well established and important risk factor for many systemic conditions, including obesity, sleep disturbance, and chronic diseases . In addition to the general health conditions, oral diseases have also been associated with depression . Although some biomarkers were reported to be associated with depression, such as inflammatory cytokines, the serum level of neurotropic factors, and the hypothalamic-pituitary-adrenal (HPA) axis hormone, the clinical use are still unclear.

In the last years, most studies have drawn attention to a contribution of depression to poor oral health status . Conversely, there are researchers investigating a possible influence of oral health conditions on depression suggesting a bi-directional relationship between oral health and mental disorders. Therefore, it can be hypothesized that treatment of periodontitis may lead to improvement in the depression score in patients.

Only few cross-sectional studies have been conducted evaluating association of depression and periodontitis that too in high income countries (Finland, USA and Korea) and the results are inconclusive. So the present study will be conducted in our country to evaluate association of periodontitis and depression to provide high level of evidence.

STUDY DESIGN AND SETTINGS The present cross sectional study will be conducted in the department of Periodontology , PGIDS, Rohtak in collaboration with the department of Psychiatry, PGIMS, Rohtak. This will be an observational cross sectional study.

STUDY PERIOD February 2020 to April 2021

METHOD OF RECRUITMENT Patients in test groups will be recruited from the Outpatient Department of Psychiatry, Post Graduate Institute of Medical Sciences, Rohtak. Patients in control group will be recruited from Department of Oral Medicine and Radiology, Post Graduate Institute of Dental Sciences, Rohtak.

BLINDING/MASKING Single blinding will be adopted where the operator assessing the periodontal parameters will be unaware regarding which group the patient belongs.

PERIODONTAL PARAMETERS :- Indices will be taken at baseline. These will be:- Plaque index Gingival index Probing pocket depth Clinical attachment loss Bleeding on probing

ELIGIBILITY:
Inclusion Criteria:

* Patients with age 18-50 years
* Newly diagnosed patients of clinical depression (international classification of diseases, classification of Mental and Behavioural Disorders, 10th Revision, Diagnostic criteria for Research35 )
* Having ≥20 natural teeth

Exclusion criteria

* Systemic disease or condition that is reported to be associated with periodontal disease, including diabetes mellitus, osteoporosis, rheumatoid arthritis, chronic renal failure, cardiovascular disease, and pregnancy
* Treatment with the following drugs in the previous 3 months: antibiotics, anti-inflammatories, steroids, immune-suppressants, lipid-lowering drugs, anticoagulants, bisphosphonates, and host modulatory drugs
* Psychiatric disorder other than depression or any other comorbid psychiatric disorder (organic mental disorder, disorders as a result of psychoactive substance use, schizophrenia and schizoaffective disorder, delirium, delusion, dementia, eating disorders, type 1 or 2 bipolar disorder, neurotic disorder, and psychotic depression)
* Treatment with any antidepressant drug
* Non-surgical or surgical periodontal treatment within the past 6 months before inclusion into the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: the study patients having mild and moderate depression as well as systemically healthy will be included .
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
clinical attachment loss | 1 year
  It will be measured from cemento-enamel junction to base of the pocket.

SECONDARY OUTCOMES:
pocket depth | 1 year
  it will be measured from gingival margin to the base of the pocket

CONTACTS AND LOCATIONS:
Overall Officials: APARNA KAUSHIK, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India